CLINICAL TRIAL: NCT06838676
Title: A Phase II Trial of ACT001 in Children and Adolescents With Diffuse Intrinsic Pontine Gliomas and H3K27-altered High Grade Gliomas
Brief Title: ACT001 for the Treatment of Diffuse Intrinsic Pontine Gliomas and H3K27-altered High Grade Gliomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Accendatech USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT2110
Record Dates: First submitted 2025-02-19; First posted 2025-02-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-02

CONDITIONS: Diffuse Intrinsic Pontine Gliomas (DIPG); Progressive DIPG; Refractory DIPG; Recurrent DIPG; H3K27-altered High Grade Glioma
Keywords: High Grade Glioma; Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma | interventions — ACT001

STUDY DESIGN:
Intervention Model Description: ACT001
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Patients with newly-diagnosed DIPG with typical MRI findings
  Interventions: Drug: ACT001
- Cohort B (Experimental): Patients with progressive/refractory/recurrent DIPG or extra-pontine H3K27-altered HGG tumors that have progressed following frontline treatment
  Interventions: Drug: ACT001

INTERVENTIONS:
Drug: ACT001 — PO BID at 875 mg/m2 for 28 days

SUMMARY:
This is a Phase II open-label study to investigate the safety and efficacy of ACT001 in patients with DIPG and H3K27-altered HGG.

DETAILED DESCRIPTION:
Patients will be enrolled on either Cohort A for newly diagnosed DIPG or on Cohort B for those with progressive / refractory DIPG or progressive / recurrent / refractory H3K27-altered HGG. Each cohort will receive ACT001 at 875 mg/m2 orally BID for 28 days (1 cycle of treatment), up to a maximum dose of 1700 mg BID. If patients are experiencing clinical benefit from study therapy, they will continue to receive ACT001 in repeat 28-day cycles for up to 26 cycles (approximately 2 years) or until disease progression, whichever occurs first. Continuation of treatment beyond 26 cycles may be considered if patients are receiving clinical benefit from the study, at the discretion of the sponsor and treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 12 months and ≤ 39 years of age at the time of study enrollment.
2. Diagnosis:

   * Cohort A: Newly Diagnosed DIPG

     * Patients with newly-diagnosed DIPG with typical MRI findings (tumors with a pontine epicenter and diffuse involvement of at least 2/3 of the pons) with or without biopsy and have completed radiation therapy (RT) within 28 to 35 calendar day prior to start of therapy.
     * Patients must have started RT <42 calendar days of radiographic diagnosis (for non-biopsied DIPG patients only) or definitive surgery, whichever is later. It is strongly recommended patients begin RT within 31 days of diagnosis/definitive surgery.

       * If a biopsy was performed, the date of surgical biopsy will be considered the date of definitive diagnostic surgery; if a patient underwent two upfront surgeries [e.g., biopsy then debulking], this is the date of the second surgery)
     * Patients must have received RT, but no other anti-cancer therapy other than surgery, and/or steroids prior to enrollment.
   * Cohort B: progressive/refractory/recurrent DIPG or H3K27-altered HGG

     * Patients with DIPG (no biopsy required) or pathologically-confirmed (at diagnosis or recurrence) extra-pontine H3K27-altered HGG who have progressive, refractory or recurrent disease following frontline treatment that included at least focal RT. Patients with refractory disease must have completed RT >6 months prior to study enrollment.
     * Patients with progressive disease only at the primary site(s) must have completed RT more than 3 months prior to enrollment.
     * Patients with progressive disease only at the primary site(s) who completed radiation therapy 3 to 6 months prior to enrollment must have had at least one follow up MRI to confirm progression (rather than pseudo- progression)
     * Patients with progressive disease due to the development a new metastatic site are eligible as long as eligibility criteria 3 (disease status) and 5 (prior RT) are met.
     * Patients with metastatic disease are eligible.
3. Disease Status

   * Cohort A: patients may have any disease status but must have completed initial radiation therapy (RT) before enrollment.
   * Cohort B: Patients must have measurable disease assessable by MRI imaging. Patients may have metastatic disease. Lesions irradiated within the last 6 months are not considered measurable unless they show definitive progression following RT.
4. Performance Level: Karnofsky Performance Scale score ≥ 50% for patients > 16 years of age and Lansky Performance Scale score > 50% for patients ≤ 16 years of age (applies to all patients) Note: Patients who are unable to walk because of paralysis, but who are capable of using a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
5. Prior anti-cancer therapy:

   * For Cohort A ONLY:
   * Patients must not have received any prior therapy other than surgery, radiation (focal to disease) and/or steroids (dexamethasone with goal to wean dexamethasone throughout protocol therapy).
   * Patients must enroll and start treatment on study between 28 and 35 calendar days post-completion of RT.
   * Patients must have started RT <42 calendar days of initial diagnosis (defined as the date of diagnostic biopsy or resection; if a patient underwent two upfront surgeries [e.g., biopsy then resection or debulking], this is the date of the second surgery).
   * Radiotherapy must have been administered at standard dose of 54 Gy for DIPG patients. Any variances in the radiotherapy dose within 10% of the standard doses outlined above will be discussed with the Study Chair (or their delegate) to confirm eligibility prior to study enrollment.
   * For Cohort B ONLY: Patients must have fully recovered from adverse events due to prior treatment with investigational or conventional agents must have recovered to a severity of Grade 0 or Grade 1 (per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or higher), with the exception of alopecia.

   Notes to the above for Cohort B: Patients with chronic Grade 2 toxicities may be eligible per discretion of the Investigator and Sponsor (e.g., Grade 2 chemotherapy-induced neuropathy). Grade 2 or 3 toxicities from prior anti-tumor therapy that are considered irreversible - defined as having been present and stable for > 6 months (such as ifosfamide-related proteinuria) may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the Investigator and Sponsor.)

   The wash out period between the prior anti-cancer chemotherapy, and first dose of ACT001 (cycle 1 day 1) must be:
   1. Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
   2. Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor.
   3. Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
   4. Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.
   5. Monoclonal antibodies: > 21 days must have elapsed from the infusion of last dose of antibody and toxicity related to antibody therapy must be recovered to Grade ≤ 1
   6. Radiation therapy:

      * For Cohort B, patients with refractory disease must have received their last fraction of frontline craniospinal or focal RT > 6 months prior to study enrollment. Patients that have received re-irradiation for progression must have received their last fraction of focal radiation >6 weeks or craniospinal radiation >6 weeks prior to study enrollment.
   7. Stem Cell Transplant: Patients must be ≥ 3 months since autologous stem cell transplant. Patients who received allogenic stem cell transplant or solid organ transplant are not eligible for study
6. Organ Function Requirements (applies to all patients)

   1. Adequate bone marrow function defined as:

      * Peripheral absolute neutrophil count (ANC) > 1000/mm³
      * Platelet count > 100,000/mm³ (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
   2. Adequate renal function defined as:

      * Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m² or
      * A serum creatinine based on age/gender as follows (Schwartz et al. J. Peds, 106:522, 1985): Age Maximum Serum Creatinine (mg/dL) Male Female 1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1.0 1.0 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4 ≥ 16 years 1.7 1.4
   3. Adequate liver function defined as:

      * total bilirubin within normal institutional limits
      * AST (serum glutamic-oxaloacetic transaminase [SGOT]) / ALT (serum glutamic-oxaloacetic transaminase [SGPT]) ≤ 2.5 × institutional upper limit of normal
      * Serum albumin ≥ 2 g/dL
   4. Adequate cardiac function defined as:

      * Ejection fraction of ≥ 50% by echocardiogram
      * QTc ≤ 480 msec (by Bazett formula)
   5. For Cohort B: Adequate neurologic function defined as:

      * Patients with seizure disorders may be enrolled if seizures are well- controlled. Well controlled is defined by no increase in seizure frequency in the 7 days prior to enrollment.
      * Patients with neurological deficits should have deficits that are stable for at least the 7 days prior to enrollment.
7. Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
8. Absence of other clinically significant concomitant active medical disorder, based on the investigator's judgement.

Exclusion Criteria:

A patient who meets any of the following exclusion criteria will not be eligible in the study (Applies to both cohorts except where noted below):

1. Cohort A only: Patients with metastatic disease.
2. Concomitant medications:

   * Corticosteroids:

     * Cohort A - Patients receiving corticosteroids are eligible regardless of dosing
     * Cohort B - Patients receiving corticosteroids who have been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are eligible
   * Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible (Refer study inclusion criteria relating to anti-cancer therapies)

     * Cohort A - Patients that have received any anti-cancer treatment other than RT are not eligible.
   * Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.
   * Anticonvulsants should be used as clinically indicated. The use of enzyme inducing anticonvulsants is not permitted
   * LHRH agonist / antagonists are not permitted
   * High Dose Biotin (B7) supplements are not permitted
3. Concomitant medications used with caution: selective serotonin reuptake inhibitor (SSRI) such as Lexapro, Fluoxetine (Prozac), fluvoxamine (Luvox), paroxetine (Paxil), sertraline (Zoloft), citalopram (Celexa), and escitalopram should be used with caution.
4. Infection: Patients who currently have an uncontrolled infection (in the opinion of the PI) are not eligible.
5. Patients who have received a prior solid organ transplantation are not eligible.
6. Pregnant or breast-feeding women will not be entered on this study due to unknown risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are postmenarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
7. Patients of childbearing or child fathering potential must agree to use adequate contraceptive methods (hormonal or barrier method of birth control; abstinence) while being treated on this study and for 3 months after completing therapy. Note: The definition of effective contraception will be based on the judgement of the principal investigator or a designated associate.
8. Patients who are in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
9. Patients who have previously received either ACT001 or parthenolide are not eligible.

Ages: 12 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2035-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) for newly diagnosed DIPG | From date on treatment until date of death due to any cause or date of last follow-up, assessed up to 60 months
  To assess the overall survival for newly-diagnosed patients with DIPG treated with RT followed by ACT001.
Objective Response Rate (ORR) in Progressive/Refractory/Recurrent HGG after frontline RT | Date on treatment through 30 days following end of protocol treatment
  To assess the rate of objective response rate (defined as partial response + complete response) in patients who have been treated with at least frontline focal RT and have progressive DIPG or progressive/recurrent/refractory H3K27-altered HGG who are treated with ACT001

SECONDARY OUTCOMES:
Overall Survival in Progressive/Refractory/Recurrent DIPG and H3K27-altered DIPG | From date on treatment until date of death due to any cause or date of last follow-up, assessed up to 60 months
  To estimate the overall survival and duration of disease control for patients who have been treated with at least RT and have progressive DIPG or progressive/recurrent/refractory H3K27-altered HGG who are treated with ACT001

CONTACTS AND LOCATIONS:
Overall Officials: David S. Ziegler, MD, FRACP, Study Chair — Sydney Children's Hospitals Network; Sara Khan, MD, PhD, FRACP, Study Chair — Nationwide Children's Hospital; Peter de Blank, MD, MSCE, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (19):
- United States (11):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Emory University/Children's Healthcare of Atlanta, Atlanta, Georgia
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philidelphia, Philidelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (2):
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Hopp Children's Cancer Center at NCT Heidelberg (KiTZ), Heidelberg, Baden-Wurttemberg, Germany
- Starship Children's Hospital, Auckland, Grafton, New Zealand

IPD SHARING:
Plan to Share IPD: No